CLINICAL TRIAL: NCT07305662
Title: Exploring the Effects of Korean-Style Mediterranean Diet (KORMED) and Physical Activity Measurement in Patients With MGUS/SMM: A Pilot Study
Acronym: KORMED-PA Stud
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo-Mee Bang, Professor, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B-2512-1017-002
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Smoldering Myeloma
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KORMED Diet and Physical Activity Monitoring (Experimental): Participants in this single-arm study will receive a 12-week Korean-style Mediterranean diet (KORMED) intervention designed to increase consumption of vegetables, fruits, whole grains, fish, legumes, and healthy oils while limiting refined carbohydrates and red or processed meats. Participants will also undergo continuous physical activity monitoring using a wearable device to measure daily step counts throughout the intervention and follow-up period. Nutritional counseling will be provided at scheduled visits (baseline, 6 weeks, and 12 weeks), and remote check-ins will support adherence. After the 12-week intervention, participants will be followed through 52 weeks to assess changes in diet adherence, physical activity, metabolic and inflammatory biomarkers, gut microbiome diversity, and quality-of-life outcomes.
  Interventions: Behavioral: KORMED Diet and Physical Activity Monitoring

INTERVENTIONS:
Behavioral: KORMED Diet and Physical Activity Monitoring — 1. KORMED Diet (Dietary Intervention) Participants will follow a Korean-style Mediterranean diet for 12 weeks. The intervention emphasizes increased intake of vegetables, fruits, legumes, whole grains, seafood, nuts, and healthy plant oils while limiting refined carbohydrates, red and processed meats, and sugar-sweetened foods. Participants receive structured dietary counseling at baseline, week 6, and week 12, with remote guidance to support adherence throughout the intervention period.
  2. Physical Activity Monitoring (Behavioral Intervention) Participants will wear an activity-tracking device throughout the 12-week intervention and subsequent follow-up. The device records daily step counts and physical activity patterns. Participants are encouraged to maintain or gradually increase daily activity, and step count feedback is reviewed during structured visits.

SUMMARY:
This single-arm pilot study aims to evaluate the feasibility and potential health effects of a Korean-style Mediterranean diet (KORMED) and continuous physical activity measurement in patients with monoclonal gammopathy of undetermined significance (MGUS) or smoldering multiple myeloma (SMM). The study investigates whether a 12-week KORMED dietary intervention, combined with monitoring of daily step counts using a wearable device, can improve metabolic and inflammatory biomarkers, body composition, gut microbiome diversity, and quality of life.

The study seeks to answer the following primary question:

Is the KORMED diet feasible and achievable for MGUS/SMM patients, as measured by changes in K-MEDAS adherence scores over 12 weeks?

Secondary questions include:

1. Does adherence to KORMED lead to improvements in BMI, inflammatory markers (CRP, IL-6), metabolic indicators (HOMA-IR, FLI), M-protein levels, and gut microbiome diversity?
2. Is increased daily physical activity, measured by step counts, associated with favorable changes in metabolic and clinical parameters?
3. Can combined dietary and activity-based lifestyle modification provide preliminary evidence supporting delayed disease progression in precursor plasma cell disorders?

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following:

Adults aged 19 to 80 years at the time of enrollment.

Diagnosed with MGUS (Monoclonal Gammopathy of Undetermined Significance) or Smoldering Multiple Myeloma (SMM) according to standard criteria.

Able and willing to follow a Korean-style Mediterranean diet (KORMED) for 12 weeks.

Able to use a smartphone and wearable device to track daily physical activity.

Willing to attend study visits and provide blood, stool, and questionnaire data at scheduled time points.

Able to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Participants will not be eligible if they meet any of the following:

Diagnosis of active multiple myeloma requiring treatment.

Current participation in another interventional clinical trial.

Severe liver, kidney, or heart disease that would make the diet or study procedures unsafe.

Uncontrolled infection or serious medical condition that may interfere with participation.

History of major gastrointestinal surgery that prevents adherence to the diet.

Pregnant or breastfeeding, or planning to become pregnant during the study period.

Allergy or intolerance to key components of the KORMED diet (e.g., fish, nuts, legumes) that prevents safe participation.

Any condition, in the investigator's judgment, that would make participation unsafe or limit the ability to complete the study.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in K-MEDAS Score From Baseline to 12 Weeks | Baseline, 12 weeks
  The primary outcome is the change in adherence to the Korean-style Mediterranean diet measured using the validated K-MEDAS questionnaire. Higher scores indicate greater diet adherence. The mean change from baseline to week 12 will be assessed.

SECONDARY OUTCOMES:
Change in Body Mass Index (BMI) From Baseline to 52 Weeks | Baseline, 6 weeks, 12 weeks, 24 weeks, 52 weeks
  BMI (kg/m²) will be measured to evaluate changes in body composition during and after the dietary intervention.
Change in Monoclonal Protein (M-protein) Levels From Baseline to 52 Weeks | Baseline, 12 weeks, 24 weeks, 52 weeks
  Serum M-protein will be quantified to explore potential effects of lifestyle intervention on clonal plasma cell activity.
Change in C-Reactive Protein (CRP), Interleukin-6 (IL-6), HOMA-IR (Insulin Resistance Index), and Fatty Liver Index (FLI) From Baseline to 52 Weeks | Baseline, 12 weeks, 24 weeks, 52 weeks
  Thsese will be measured to evaluate inflammatory response to the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) due to privacy considerations and institutional restrictions. Only aggregated results will be shared in publications